CLINICAL TRIAL: NCT06951139
Title: The Effect of Molar Incisor Hypomineralisation on the Stomatognathic System in Children: A Prospective Study
Brief Title: The Effect of Molar Incisor Hypomineralisation on the Stomatognathic System
Status: Completed | Type: Observational
Sponsor: Ozge Gungor (Other)
Responsible Party: Sponsor-Investigator, Ozge Gungor, PhD, DDS, Assoc. Prof. Dr., Akdeniz University
Organization: Akdeniz University (Other)
Other Study IDs: TBAEK-75
Record Dates: First submitted 2025-03-28; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Molar Incisor Hypomineralization
Keywords: elasticity; temporomandibular disorders; ultrasound; masticatory muscle
MeSH Terms: conditions — Molar Hypomineralization; Temporomandibular Joint Disorders | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- MIH Group: This group includes children aged 9-14 years diagnosed with Molar Incisor Hypomineralization (MIH). Participants in this group underwent clinical and ultrasonographic evaluation to assess temporomandibular joint function and masticatory muscle properties.
  Interventions: Diagnostic Test: Ultrasound and Shear Wave Elastography
- Control Group: This group includes healthy children aged 9-14 years without a diagnosis of Molar Incisor Hypomineralization (MIH). Participants were evaluated using the same clinical and ultrasonographic procedures as the MIH group.
  Interventions: Diagnostic Test: Ultrasound and Shear Wave Elastography

INTERVENTIONS:
Diagnostic Test: Ultrasound and Shear Wave Elastography — Non-invasive diagnostic imaging techniques used to assess the stomatognathic system. Ultrasound was performed to measure the thickness of the masseter, temporalis, and sternocleidomastoid muscles, as well as the articular disc of the temporomandibular joint. Shear Wave Elastography was used to evaluate the elasticity (stiffness) of the same muscles and joint structures in kilopascals. All evaluations were conducted at rest, using standardized positioning, and by the same experienced operator.

SUMMARY:
This study aims to examine whether children with Molar Incisor Hypomineralization (MIH) are more likely to have problems with the jaw joint and chewing muscles. MIH is a dental condition where the enamel of the first molars and incisors is weaker than normal. The researchers performed clinical examinations and ultrasound imaging to evaluate the thickness and elasticity of the chewing muscles. They also used a questionnaire to check for symptoms of temporomandibular disorders (TMD), such as jaw pain, headaches, and joint sounds.

DETAILED DESCRIPTION:
This prospective clinical study investigates the potential impact of Molar Incisor Hypomineralization (MIH) on the stomatognathic system in children. MIH is a developmental enamel defect that affects the first permanent molars and incisors, resulting in weakened enamel and increased sensitivity. While MIH has been well documented in the context of dental health, its broader functional consequences remain underexplored. A total of 84 children aged 9-14 years participated in this study, including 43 with MIH and 41 healthy controls. The evaluation involved both clinical and ultrasonographic examinations. Temporomandibular disorders (TMD) were assessed using the Fonseca Anamnestic Index and through clinical parameters such as joint sounds, headaches, mandibular deviation/deflection, and mouth opening limitation. Ultrasound imaging, including shear wave elastography, was used to evaluate the thickness and elasticity of the masseter, temporalis, and sternocleidomastoid muscles, as well as the articular disc of the temporomandibular joint.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 9 and 14 years
* Good general health with no systemic disease
* Score of 3 or 4 on the Frankl Behavior Rating Scale
* No parafunctional oral habits (e.g., bruxism)
* No skeletal orthodontic abnormalities
* For the MIH group: presence of at least one first permanent molar diagnosed with MIH
* For the control group: absence of MIH diagnosis

Exclusion Criteria:

* Presence of advanced periodontal disease or tooth mobility
* History of facial trauma or jaw fracture
* Current medication use
* Inability to cooperate during clinical or ultrasonographic examinations
* Any condition that may affect temporomandibular joint structure or function

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children aged 9 to 14 years who visited the pediatric dentistry clinic for routine examinations. The study included both children diagnosed with Molar Incisor Hypomineralization (MIH) and healthy controls without MIH.
Sampling Method: Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2025-03-20 (Actual)

PRIMARY OUTCOMES:
Prevalence of temporomandibular disorders (TMD) in children with MIH | At the time of enrollment (single clinical visit)
  The presence of TMD was assessed in both the MIH and control groups using the Fonseca Anamnestic Index and clinical examination. TMD diagnosis was based on signs such as joint sounds, deviation/deflection, headaches, and mouth opening limitation.
Thickness of masticatory muscles in children with and without MIH | At the time of enrollment (single clinical visit)
  Ultrasound and shear wave elastography were used to evaluate the thickness (in millimeters) of the masseter, temporalis, and sternocleidomastoid muscles bilaterally in both groups. Mean values were calculated and compared.
Elasticity of masticatory muscles in children with and without MIH | At the time of enrollment (single clinical visit)
  Ultrasound and shear wave elastography were used to evaluate the elasticity (in kilopascals) of the masseter, temporalis, and sternocleidomastoid muscles bilaterally in both groups. Mean values were calculated and compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University Faculty of Dentistry, Department of Pediatric Dentistry, Antalya, Konyaaltı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No